CLINICAL TRIAL: NCT05488925
Title: Comparison of Preoperative Analgesics on the Efficacy of Inferior Alveolar Nerve Block on Patients With Symptomatic Irreversible Pulpitis: a Double Blinded, Randomized Controlled Trial.
Brief Title: Comparison of Preoperative Analgesics on the Efficacy of Inferior Alveolar Nerve Block.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Farjad Zafar (Other)
Responsible Party: Sponsor-Investigator, Farjad Zafar, Assistant Professor and Head of Department of Dental Implantology, Baqai Medical University
Organization: Baqai Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BDC/ERB/2021/016
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: inferior alveolar nerve block; irreversible pulpitis; diclofenac sodium; piroxicam; tramadol
MeSH Terms: interventions — Vitamin E; Diclofenac; Piroxicam; Tramadol

STUDY DESIGN:
Intervention Model Description: The visual analogue scale was used to assess the patients' pain levels prior to the drug ingestion. The patients were then given their respective group of drug where the control group received vitamin E and three experimental groups received one tablet/capsule of diclofenac sodium (Voltral SR100, 100 mg), piroxicam (Feldene, 20 mg), and tramadol (Tramal, 50 mg). The patients were instructed to wait for 1 hour before they were administered an inferior alveolar nerve block. Standard root canal treatment was initiated after lip numbness was achieved, and pain levels were reassessed by visual analogue scale.
Who Masked: Participant, Care Provider
Masking Description: The study was designed to be a double blinded study, where the operators and the patients both were unaware of the groups of drugs that were used; this anonymity was achieved by marking the groups A, B, C and D on boxes for drugs containing a placebo, diclofenac sodium, piroxicam, and tramadol respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Vitamin E (Placebo Comparator)
  Interventions: Drug: Vitamin E
- Diclofenac sodium (Experimental)
  Interventions: Drug: Diclofenac Sodium
- Piroxicam (Experimental)
  Interventions: Drug: Piroxicam
- Tramadol (Experimental)
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Vitamin E — Evion, 400 mg
  Arms: Vitamin E
Drug: Diclofenac Sodium — Voltral SR100, 100 mg
  Arms: Diclofenac sodium
Drug: Piroxicam — Feldene, 20 mg
  Arms: Piroxicam
Drug: Tramadol — Tramal, 50 mg
  Arms: Tramadol

SUMMARY:
The purpose of this study is to see how preoperative oral diclofenac sodium, piroxicam, and tramadol affects inferior alveolar nerve block efficacy during root canal treatment of mandibular molars with symptomatic irreversible pulpitis.

The proposed hypothesis is that the tested drug groups will improve the efficacy of inferior alveolar nerve block in comparison to the control group.

DETAILED DESCRIPTION:
Standard Operating Procedure:

* A non-probability consecutive sampling was done in a dental out patient department and 120 patients were included and randomly divided in the 4 groups (n=30) using simple randomization as per the inclusion criteria.
* A verbal informed consent was taken from each participant before including them in a group.
* The study was designed to be a double blinded study, where the researchers and the patients both were unaware of the groups of drugs that were used; this anonymity was achieved by marking the groups A, B, C and D on boxes for drugs containing a placebo, diclofenac sodium, piroxicam, and tramadol respectively.
* The Heft Parker Visual Analogue Scale was used to assess the patients' pain levels prior to the drug ingestion, and the study was continued on the patients that reported moderate to severe pain on the Visual Analogue Scale. On this scale, the pain intensities were categorized as: no pain (0), mild pain (1-54 mm), moderate pain (55- 114 mm) and severe pain (> 114 mm).
* The patients were then given their respective group of drug/placebo. The patients were instructed to wait for 1 hour before they were administered Inferior Alveolar Nerve Block with 1.8 ml of 2% lidocaine with 1:100000 epinephrine using a non-aspirating syringe through a long needle of 27-Gauge.
* Standard root canal treatment was initiated after lip numbness was achieved, and pain levels were reassessed by Heft Parker Visual Analogue Scale during the root canal procedure. However, the patients who did not achieve the numbness of the lips were excluded from the study.
* Patients who reported discomfort and pain during the endodontic procedure were intervened appropriately; conversely, if the patient did not report any intraoperative pain, endodontic procedure was resumed.
* Till the end of the data collection process, the collected data forms were stored in a 4 different files labeled A ,B ,C and D respective to the drug groups. On completion of the collection process the data was added and stored as a data file into IBM SPSS Statistics version 25 and further analyzed.

Sample Size Estimation:

The study size was calculated with reference to previous reports, revealing that at least 30 individuals should be included as per the analysis of power of the study. The value of power used was 0.96, the effect size was taken as 0.4, and α was set as 0.05.

Statistical Analysis Plan:

Test of normality will be checked using one sample Shapiro Wilk. One-way ANOVA with Tukey's post-hoc will be employed if parametric test criteria is met; however if the parametric criteria is not fulfilled, the experimental groups will be compared using Kruskal-Wallis test with post-hoc analysis. The Chi-square test will be used to compare gender and drug groups against the Inferior Alveolar Nerve Block efficacy. These tests will be conducted on SPSS Statistics version 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 - 65 years.
* Patients with no medical or systemic conditions.
* Patients with prolonged pain response on cold pulp testing of 1st and 2nd mandibular molars.
* Patient with 1st and 2nd mandibular molars having symptomatic irreversible pulpitis with no periapical pathology or tenderness on percussion.
* Preoperative moderate to severe pain on heft parker visual analogue scale.
* Patients who can understand the recording of the pain using heft parker visual analogue scale.

Exclusion Criteria:

* Patients who are pregnant and/or breastfeeding.
* Patients with reported allergy to diclofenac sodium, piroxicam, and tramadol.
* Patients with periodontal pathologies, necrotized pulp, ankylosed or resorbed roots, open apex and non-restorable tooth.
* Patients who have taken an analgesic in the past 24 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
To check the efficacy of preoperative analgesics on inferior alveolar nerve block using Heft-Parker Visual Analogue Scale. | 1 hour
  Study's outcome is to evaluate the efficacy of different preoperative oral analgesics on inferior alveolar nerve block during root canal procedure of mandibular teeth using Heft-Parker Visual Analogue Scale on symptomatic irreversible pulpitis patients
  Heft-Parker Visual Analogue Scale is a visual assessment tool to record patients pain intensity. This scale is categorized as: no pain (0mm), moderate pain (55-114mm), and severe pain (>114mm)
  * Patients will register their Heft-Parker Visual Analogue Scale recording to the investigator before drug ingestion
  * Patients will re-register their Heft-Parker Visual Analogue Scale 1 hour after the drug ingestion, during root canal procedure after inferior alveolar nerve block
  * The difference in the preoperative and intraoperative Heft-Parker Visual Analogue Scale score will determine the efficacy of different analgesic interventional groups

CONTACTS AND LOCATIONS:
Overall Officials: Farjad Zafar, BDS, MSc, Study Director — Assistant Professor and Head of Department of Dental Implantology.; Maryam Riaz, BDS, Principal Investigator — Lecturer in Department of Oral Biology.; Zara Khalid, BDS, Principal Investigator — House officer.; Tipu Sultan, BDS, MDS, Principal Investigator — Assistant Professor in Department of Periodontology.; Aisha Wali, BDS, MPH, Study Director — Assistant Professor and Head of Department of Research and Development.; Talha M Siddiqui, BDS, MCPS, Study Chair — Professor and Chairman of Operative Dentistry and Endodontics.
Locations (1):
- Department of Operative Dentistry, Baqai Dental College, Baqai Medical University., Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared with the researchers who have received an ethical approval from their institution/organization through an email.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available by November 2022 and will be available for 5 years till October 2027.
Access Criteria: Researchers who have received an ethical approval from their institution/organization will be provided with the collected IPD.
  The data will be sent through an email.

REFERENCES:
- [Result] Prasanna N, Subbarao CV, Gutmann JL. The efficacy of pre-operative oral medication of lornoxicam and diclofenac potassium on the success of inferior alveolar nerve block in patients with irreversible pulpitis: a double-blind, randomised controlled clinical trial. Int Endod J. 2011 Apr;44(4):330-6. doi: 10.1111/j.1365-2591.2010.01833.x. PMID 21692235

DOCUMENTS (2):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05488925/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05488925/SAP_001.pdf